CLINICAL TRIAL: NCT01748110
Title: Health Interventions in Men Undergoing Radical Prostatectomy- A Randomized Controlled Clinical Trial
Brief Title: Health Interventions in Men Undergoing Radical Prostatectomy
Acronym: HIM-UP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding could not be secured
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NA_00070555
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Prostate Cancer; Erectile Dysfunction Following Radical Prostatectomy; Urinary Incontinence
Keywords: quality of life; erectile function
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Local Control Group (No Intervention): This arm is for patients in the District of Columbia (DC), (Maryland) MD, (Virginia) VA area that are able to attend all follow up visits at 3 month, 6 month, 12 month and 18 months post operative periods that have been randomized to standard recommendations for fitness/health interventions prior to surgery.
- Local TRIMM Group (Experimental): This arm is for patients in the DC, MD, VA area that are able to attend all follow up visits at 3 month, 6 month, 12 month and 18 months post operative periods that have been randomized to receive daily text message reminder and prompts targeted to the patient's dietary, fitness and urologic goals and needs using the Tailored Rapid Interactive Mobile Messaging (TRIMM) method. Patients will receive these text messages from 4 weeks prior to surgery until 8 week after surgery
  Interventions: Behavioral: TRIMM
- Local Intensive Group (Experimental): This arm is for patients in the DC, MD, VA area that are able to attend all follow up visits at 3 month, 6 month, 12 month and 18 months post operative periods that have been randomized to undergo intensive in-person fitness interventions according to the Look AHEAD model. This will involve attendance at weekly support group meetings and personal monthly meetings with a health care provider/
  Interventions: Behavioral: Intensive Fitness Intervention
- Distant Control Group (No Intervention): This arm is for geographically distant patients that are unable to attend all follow up visits at 3 month, 6 month, 12 month and 18 months post operative periods that have been randomized to standard recommendations for fitness/health interventions prior to surgery.
- Distant TRIMM Group (Experimental): This arm is for geographically distant patients that are unable to attend all follow up visits at 3 month, 6 month, 12 month and 18 months post operative periods that have been randomized to receive daily text message reminder and prompts targeted to the patient's dietary, fitness and urologic goals and needs using the Tailored Rapid Interactive Mobile Messaging (TRIMM) method. Patients will receive these text messages from 4 weeks prior to surgery until 8 week after surgery
  Interventions: Behavioral: TRIMM

INTERVENTIONS:
Behavioral: Intensive Fitness Intervention — This intervention will involve adhering to health interventions such as behavior and diet modification, and exercise. Patients will follow-up monthly with a health counselor to verify progress.
  Other Names: Look AHEAD model
  Arms: Local Intensive Group
Behavioral: TRIMM — text message intervention.
  Other Names: Tailored Rapid Interactive Mobile Messaging
  Arms: Distant TRIMM Group; Local TRIMM Group

SUMMARY:
The goal of the study is to assess the impact of a health intervention, involving both diet and exercise modification, on outcomes following radical prostatectomy for the treatment of clinically localized prostate cancer. The specific urological outcomes expected to be improved are accelerated and/or improved recovery of erectile function (EF), as well as urinary continence, both very commonly affected by this surgery. Furthermore, as demonstrated by changes in responses to various questionnaires, an improvement in overall health-related quality of life is expected. Finally, an improvement in patients participating in the intervention groups in physical parameters, including body mass index (BMI), blood pressure (BP), and metabolic parameters, including serum glucose and cholesterol levels, is expected.

DETAILED DESCRIPTION:
This project will assess whether a health-promotion intervention initiated prior to and continuing beyond radical prostatectomy for the treatment of clinically localized prostate cancer results in improvements in overall health, health-related quality of life, and specific urological outcomes, specifically recovery of EF and urinary continence. While there is an abundance of literature supporting the harmful impact that obesity has on prostate cancer risk, delayed diagnosis, surgical outcomes, pathological outcomes and overall mortality, there is a paucity of data on the impact of health/fitness interventions on immediate post-operative quality of life outcomes.

Data supporting the benefit of lifestyle interventions in terms of overall health come from the Look AHEAD trial [1], which demonstrated clinically significant weight loss and improvements in diabetic control and cardiovascular risk factors in obese, type 2 diabetics. It is expected that this intervention will result in beneficial changes to the participants' overall health status as represented in the short term by improvements in objective clinical measurements (such as reduction in weight, BP, serum cholesterol and fasting serum glucose levels), and overall health-related quality of life. The investigators also hypothesize that such an intervention will result in improved post-operative urological outcomes, namely accelerated return of urinary continence and EF. Urologists are in a good position to promote healthy living, and initiating interventions such as these prior to surgery can provide the foundation of a healthy lifestyle that will enable the patient to maintain the aforementioned benefits well beyond their surgery, and extending beyond the urological domain.

The goal is to prove that patients participating in one of two lifestyle interventions, a more intense health promotion intervention or a less intense text-message program, will report improved physical parameters: BMI, BP, metabolic parameters (fasting serum glucose, serum cholesterol), health-related quality of life, recovery of EF and urinary continence (the latter three as reported by questionnaires) compared to patients who are given standard advice prior to radical prostatectomy.

Specific Aim: To evaluate by means of a randomized, controlled, clinical trial the relative benefits and costs of an intensive health-promotion intervention, compared with a less intensive intervention consisting of regular daily text message health reminders, compared with the standard advice given to patients undergoing radical prostatectomy. While it is intuitive that healthier patients will feel better and have easier recoveries after radical prostatectomy, there is no existing evidence thus far to support this. The investigation will apply a single center, randomized, clinical 18 month study design and employ validated instruments to assess health related quality of life status, EF and urinary continence.

The study design will be a single center, randomized, clinical 3-arm study, comparing the effects of an intensive lifestyle intervention based on the Look AHEAD regimen vs. a less intensive text message intervention vs. standard lifestyle advice typically provided prior to radical prostatectomy. For the control arm, participants will complete post-operative assessments at months 3, 6, 12 and 18 where they will repeat the baseline questionnaires and measures. Please note that for all recruited patients who are not local, the follow-up questionnaires will be obtained via mail, and the physical parameters will be derived from direct contact with the patient's local care provider. In the event that this is not possible, we will rely on patient self-report. Standard practice associated with surgery and postoperative laboratory testing will be performed. Patients may use a phosphodiesterase type 5 inhibitor (sildenafil, tadalafil or vardenafil) following surgery as conventional "on-demand" therapy for erectile dysfunction (ED).

For the text message (Tailored Rapid Interactive Mobile Messaging-TRIMM) arm, same as above for standard care, plus: "Push" and "pull"-type text messages will be delivered at a frequency of 3-4 times/day, starting at least 4 weeks prior to surgery and continuing 8 weeks postoperatively. Specific content has been developed and field-tested for acceptability. Patients will be asked to select three of seven possible health-related goals targeting specific categories, including dietary (such as increasing fruit and vegetable consumption), exercise (such as more walking) and behavioral (such as less eating in response to stress) goals. All text message participants will also receive semi-weekly messages related to specific urological goals relating to their surgery, such as performing Kegel exercises and maintaining intimate relationships. At least one message daily will require a response, and targeted feedback will be given based on the response. For example, participants will be issued a pedometer and asked to record their daily steps. If steps reported for the day are above or below goal, automatically generated instructions/praise/alternatives will be proffered.

For the intensive intervention, same as standard care, plus: Weekly meetings, starting at least 4 weeks prior to surgery and continuing 8 weeks postoperatively, consisting of support group meetings 3 times/month using the Look AHEAD curriculum modified to a shorter term intervention, plus a monthly individual follow-up visit. This individual monthly visit would include a focused evaluation of the participant, including review of his goals and feedback on his progress. The intensive intervention will provide both relevant diet and exercise education and support for long-term lifestyle changes. The intensive intervention will be facilitated by a physician or other trained provider. At each monthly visit, patient's weight will be recorded and a review of their activity and diet logs conducted. A topical lesson corresponding to the Look AHEAD curriculum [1] will be given and participants would be given a chance to discuss the lesson and any road-blocks to their progress that have occurred. Participants will be issued a pedometer and asked to record their daily steps, to be used as a surrogate for physical activity.

The sample size will be 25 patients randomized to each study arm. There will be a total of 5 arms (a total of 125 patients), with the study being divided based on patient proximity to the Johns Hopkins Hospital. Local patients (defined as those patients who are able to be physically present for all of the study sessions as well as follow-up appointments) will be randomized to 3 arms: control, TRIMM and intensive intervention. Distant patients (defined as patients who are not able to be present for all study sessions as well as follow-up appointments) will be randomized to 2 arms: control and TRIMM. Study procedures will involve screening and informed consent after initial consultation, baseline evaluation including medical clearance and completion of validated questionnaires. Randomization will be achieved by a computerized random number generator, with patients stratified based on age. Assessment tools will consist of the IIEF questionnaire, the Quality of Erection Questionnaire (QEQ) and health related quality of life instruments: RAND 12-item Health Survey (SF-12) and the Expanded Prostate Cancer index Composite Short Form (EPIC-26-sexual and urinary domains). Standard practice associated with surgery, blood transfusion and postoperative laboratory testing will be performed. Patients will be prescribed a phosphodiesterase type 5 inhibitor (sildenafil, tadalafil or vardenafil) at 1 month following surgery to be used as conventional "on-demand" therapy. Adverse event monitoring will be performed.

ELIGIBILITY:
Inclusion Criteria:

* men 40-65 years of age
* localized prostate cancer (clinical stage < T2b, Gleason grade < 7, pre-operative prostate specific antigen (PSA) < 10)
* scheduled to undergo curative nerve-sparing prostatectomy at the Johns Hopkins Hospital

Exclusion Criteria:

* in a stable relationship for at least 6 months
* moderately to severely impaired preoperative erectile function (IIEF-erectile function domain score < 16)
* answering less than 2-3 times or > to question #6 on the IIEF
* severe lower urinary tract symptoms International Prostate Symptom Score (IPSS) >20

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in erectile function (EF) | From baseline (4 weeks before surgery) to 3 months after surgery
  The International Index of Erectile Function (IIEF) will be administered. This is a 15 item questionnaire . The questionnaire measures Erectile Function (scored from 0-30), Intercourse satisfaction (0-15), orgasmic function (0-10), Sexual Desire (2-10) and Overall satisfaction (2-10).
Change in EF | From baseline (4 weeks before surgery) to 6 months after surgery
  The International Index of Erectile Function (IIEF) will be administered. This is a 15 item questionnaire . The questionnaire measures Erectile Function (scored from 0-30), Intercourse satisfaction (0-15), orgasmic function (0-10), Sexual Desire (2-10) and Overall satisfaction (2-10).
Change in EF | From baseline (4 weeks before surgery) to 12 months after surgery
  The International Index of Erectile Function (IIEF) will be administered. This is a 15 item questionnaire . The questionnaire measures Erectile Function (scored from 0-30), Intercourse satisfaction (0-15), orgasmic function (0-10), Sexual Desire (2-10) and Overall satisfaction (2-10).
Change in EF | From baseline (4 weeks before surgery) to 18 months after surgery
  The International Index of Erectile Function (IIEF) will be administered. This is a 15 item questionnaire . The questionnaire measures Erectile Function (scored from 0-30), Intercourse satisfaction (0-15), orgasmic function (0-10), Sexual Desire (2-10) and Overall satisfaction (2-10).
Change in EF | From baseline (4 weeks before surgery) to 3 months after surgery
  The Quality of Erection (QEL) questionnaire will be administered. This is a 6 item questionnaire addressing the patient's perception of erectile rigidity during sexual activity. It is scored from 0-100 with 100 indicating the highest quality erection
Change in EF | From baseline (4 weeks before surgery) to 6 months after surgery
  The Quality of Erection (QEL) questionnaire will be administered. This is a 6 item questionnaire addressing the patient's perception of erectile rigidity during sexual activity. It is scored from 0-100 with 100 indicating the highest quality erection
Change in EF | From baseline (4 weeks before surgery) to 12 months after surgery
  The Quality of Erection (QEL) questionnaire will be administered. This is a 6 item questionnaire addressing the patient's perception of erectile rigidity during sexual activity. It is scored from 0-100 with 100 indicating the highest quality erection
Change in EF | From baseline (4 weeks before surgery) to 18 months after surgery
  The Quality of Erection (QEL) questionnaire will be administered. This is a 6 item questionnaire addressing the patient's perception of erectile rigidity during sexual activity. It is scored from 0-100 with 100 indicating the highest quality erection
Change in Urinary function | From baseline (4 weeks before surgery) to 3 months after surgery
  The expanded prostate cancer index (EPIC-26) urinary domain will be administered. This is a 7 item questionnaire addressing the patient's perception of their urinary function over the previous 4 weeks. Higher scores indicate a greater degree of urinary dysfunction
Change in Urinary function | From baseline (4 weeks before surgery) to 6 months after surgery
  The expanded prostate cancer index (EPIC-26) urinary domain will be administered. This is a 7 item questionnaire addressing the patient's perception of their urinary function over the previous 4 weeks. Higher scores indicate a greater degree of urinary dysfunction
Change in Urinary function | From baseline (4 weeks before surgery) to 12 months after surgery
  The expanded prostate cancer index (EPIC-26) urinary domain will be administered. This is a 7 item questionnaire addressing the patient's perception of their urinary function over the previous 4 weeks. Higher scores indicate a greater degree of urinary dysfunction
change in urinary function | From baseline (4 weeks before surgery) to 18 months after surgery
  The expanded prostate cancer index (EPIC-26) urinary domain will be administered. This is a 7 item questionnaire addressing the patient's perception of their urinary function over the previous 4 weeks. Higher scores indicate a greater degree of urinary dysfunction

SECONDARY OUTCOMES:
change in health related quality of life | From baseline (4 weeks before surgery) to 3 months after surgery
  The RAND 12 questionnaire will be administered. This is a validated questionnaire evaluating the patient's perception of their overall health.
change in health related quality of life | From baseline (4 weeks before surgery) to 6 months after surgery
  The RAND 12 questionnaire will be administered. This is a validated questionnaire evaluating the patient's perception of their overall health.
change in health related quality of life | From baseline (4 weeks before surgery) to 12 months after surgery
  The RAND 12 questionnaire will be administered. This is a validated questionnaire evaluating the patient's perception of their overall health.
change in health related quality of life | From baseline (4 weeks before surgery) to 18 months after surgery
  The RAND 12 questionnaire will be administered. This is a validated questionnaire evaluating the patient's perception of their overall health.
change in sexual satisfaction | From baseline (4 weeks before surgery) to 3 months after surgery
  The EPIC-26 sexual domain questionnaire will be administered. This is a 9 item questionnaire used to evaluate the patient's perception of their sexual satisfaction over the previous 4 weeks. Higher scores indicate greater dissatisfaction and dysfunction
change in sexual satisfaction | From baseline (4 weeks before surgery) to 6 months after surgery
  The EPIC-26 sexual domain questionnaire will be administered. This is a 9 item questionnaire used to evaluate the patient's perception of their sexual satisfaction over the previous 4 weeks. Higher scores indicate greater dissatisfaction and dysfunction
change in sexual satisfaction | From baseline (4 weeks before surgery) to 12 months after surgery
  The EPIC-26 sexual domain questionnaire will be administered. This is a 9 item questionnaire used to evaluate the patient's perception of their sexual satisfaction over the previous 4 weeks. Higher scores indicate greater dissatisfaction and dysfunction
change in sexual satisfaction | From baseline (4 weeks before surgery) to 18 months after surgery
  The EPIC-26 sexual domain questionnaire will be administered. This is a 9 item questionnaire used to evaluate the patient's perception of their sexual satisfaction over the previous 4 weeks. Higher scores indicate greater dissatisfaction and dysfunction
Change in Body mass index (BMI) | From baseline (4 weeks before surgery) to 3 months after surgery
Change in Body mass index (BMI) | From baseline (4 weeks before surgery) to 6 months after surgery
Change in Body mass index (BMI) | From baseline (4 weeks before surgery) to 12 months after surgery
Change in Body mass index (BMI) | From baseline (4 weeks before surgery) to 18 months after surgery
Change in serum cholesterol level | From baseline (4 weeks before surgery) to 3 months after surgery
Change in serum cholesterol level | From baseline (4 weeks before surgery) to 6 months after surgery
Change in serum cholesterol level | From baseline (4 weeks before surgery) to 12 months after surgery
Change in serum cholesterol level | From baseline (4 weeks before surgery) to 18 months after surgery
Change in blood pressure (BP) | From baseline (4 weeks before surgery) to 3 months after surgery
Change in blood pressure (BP) | From baseline (4 weeks before surgery) to 6 months after surgery
Change in blood pressure (BP) | From baseline (4 weeks before surgery) to 12 months after surgery
Change in blood pressure (BP) | From baseline (4 weeks before surgery) to 18 months after surgery
Change in serum glucose | From baseline (4 weeks before surgery) to 3 months after surgery
Change in serum glucose | From baseline (4 weeks before surgery) to 6 months after surgery
Change in serum glucose | From baseline (4 weeks before surgery) to 12 months after surgery
Change in serum glucose | From baseline (4 weeks before surgery) to 18 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Arthur L Burnett, MD, MBA, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States